CLINICAL TRIAL: NCT02454543
Title: Multicentric, Prospective, Randomized Controlled Trial Comparing Best Systemic Therapy (BST) With Radical Prostatectomy or BST Alone in the Management of Men With Pauci-metastatic Prostate Cancer
Brief Title: Impact of Radical Prostatectomy as Primary Treatment in Patients With Prostate Cancer With Limited Bone Metastases
Acronym: g-RAMPP
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Martini-Klinik am UKE GmbH (Other)
Collaborators: Förderverein Hilfe bei Prostatakrebs e.V. (Unknown)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: G-RAMPP_MK-2014; AP 75/13 (Other: Arbeitsgemeinschaft urologische Onkologie)
Record Dates: First submitted 2015-05-08; First posted 2015-05-27 (Estimated); Last update posted 2026-01-12 (Actual); Status verified 2026-01

CONDITIONS: Prostate Cancer
Keywords: metastatic; prostatectomy; androgen deprivation; best systemic therapy
MeSH Terms: conditions — Prostatic Neoplasms; Neoplasm Metastasis | interventions — Androgen Antagonists; Drug Therapy

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Radical prostatectomy and BST (Other): BST plus radical prostatectomy with ext. lymphadenectomy
  Interventions: Procedure: Radical prostatectomy
- Best Systemic Therapy (BST) (Other): e.g. Androgen deprivation therapy, chemotherapy, others
  Interventions: Drug: Best systemic therapy

INTERVENTIONS:
Procedure: Radical prostatectomy — Study participants randomized in the intervention arm receive best systemic therapy in addition to radical prostatectomy with extended lymphadenectomy. It is not crucial whether the radical prostatectomy is performed open or robot-assisted.
  Arms: Radical prostatectomy and BST
Drug: Best systemic therapy — For the antiandrogenic therapy a non-steroidal antiandrogen (e.g. flutamide, bicalutamide) or a gonadotropin-releasing hormone (GnRH) analogues (e.g. goserelin, leuprolide) are available.
  The selection of best systemic therapy is up to the judgment of the treating urologist.
  Other Names: Androgen deprivation therapy, chemotherapy, others
  Arms: Best Systemic Therapy (BST)

SUMMARY:
The aim of the study is to investigate, the effect of radical prostatectomy with extended lymphadenectomy on cancer-specific survival, time to castration-resistance, time to progression and quality of life in patients with a limited bone metastatic prostate cancer. In addition the influence of patient- and disease-related factors on clinical outcome (prognostic effect) and on the comparison therapy (predictive effect) will be examined.

Amendment05: Due to the slow tumor biology of prostate cancer, the follow-up period of 5 years is not sufficient to reach the primary endpoint of the study. For this reason, the follow-up is extended for a further 5 years with 2 visits per year.

DETAILED DESCRIPTION:
More recent data has shown that performing local therapy with lymphogenic metastatic prostate cancer has resulted in a definite benefit in cancerspecific and overall survival. The analysis of this data has led to a change of paradigm in the treatment of lymphogenic metastatic prostate cancer (Isbarn Deutsches Ärzteblatt 2013). Patients with low lymphogenic metastatic load and low comorbidity are therefore frequently given local therapy. In a retrospective review of patients with lymphogenic metastatic prostate cancer, who were either treated by means of best systemic therapy or best systemic therapy plus radical prostatectomy, a highly significant benefit is shown for the patient group which received surgery (Engel et al., Eur Urol 2012). The 5 and 10 year overall survival rate in this cohort was 84% and 64% respectively following RP and in the other cohort with best systemic therapy without RP 60% and 28% respectively.

Our own working group was able to confirm this clear survival benefit in the lymphogenic metastatic stage for patients who received surgery: in a matched pair analysis the clinically progression-free survival rate after 5 and 10 years was 77% and 61% respectively after additional RP and 61% and 31% respectively with best systemic therapy alone (p=0.005). The same trend was found for cancer-specific survival (84% and 76% with additional RP versus 81% and 46% with best systemic therapy alone (p=0.001) (Steuber et al., BJUI 2011).

The impressive improvements in the survival rates of lymphogenic metastatic prostate cancer through local therapy compared with best systemic therapy alone suggests that patients with distant metastases could potentially also benefit from local therapy. Besides possible effects on tumour control, the RP could also be beneficial with regard to a local progression of the prostate cancer (rectal infiltration, infiltration of the bladder). This could lead to an improvement in the quality of life in the course of the disease. On the other hand, radical prostatectomy is associated with potential side-effects (e.g. urinary incontinence in approximately 5 - 10% of patients as well as possible general side-effects, such as thrombosis, embolism, impaired wound healing etc.), which can lead to a loss in terms of quality of life.

ELIGIBILITY:
Patients with locally resectable intermediate and high-risk prostate cancer which has been confirmed by biopsy according to D'Amico criteria (intermediate risk: PSA 10-20 ng/ml, cT2b-c, Gleason score 7; high risk: PSA >20 ng/ml, >cT2c, Gleason score 8-10) with clinical evidence of bone metastases in imaging tests can be included. Necessary radiotherapy of the bone metastases as required is also permitted prior to inclusion in the study.

In line with the results from the recent CHAARTED and STAMPEDE studies (Sweeny et al., 2015, James et al 2015), early treatment with taxanes may be used in both the standard treatment arm as well as in the intervention arm where the prostatektomie is performed. The period 6 months from the initial diagnosis to randomization and possibly three months from randomization to surgery must be complied with.

Inclusion criteria

1. Patients with newly diagnosed prostate cancer which has been confirmed by histological examination (within the last 6 months prior to randomization)
2. At least one and at most 5 bone metastases in imaging tests (bone scintigraphy, CT, MRT or PET) at diagnosis with no evidence of visceral metastasis. Patients with evidence of lymph node metastasis (N1) are allowed
3. PSA ≤ 200 ng/ml at diagnosis (without ADT)
4. Asymptomatic or mild symptomatic disease
5. Locally resectable tumour stage
6. ECOG Performance Score 0-1
7. Submission of the patient's written declaration of informed consent following explanation
8. Age ≥ 18 - ≤ 75 years
9. Full legal capacity and compliance of the Patient

Exclusion Criteria:

* Contraindications to radical prostatectomy (Local non-resectable disease, increased anesthetic risk due to comorbidities)
* Detection of more than 5 bone metastases
* Pain management with opioid analgetics
* Evidence of visceral metastases or brain metastases
* Neuroendocrine and / or small cell differentiation in histology of the biopsy
* Charlson Comorbidity Index > 2
* ECOG Performance Score > 1
* Myocardial infarction or stroke within the last 6 months
* Existing major cardiovascular (grade III - IV according to NYHA), pulmonary (pO2 <60 mmHg), renal, hepatic or hematopoietic disease (e.g. severe bone marrow aplasia)
* Severe psychiatric disorders persons housed on judicial or administrative arrangement in an institution
* Simultaneous participation in another clinical trial with interventional character of the metastatic prostate cancer

Ages: 18 Years to 75 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 452 (Estimated)
Dates: Start 2015-05; Primary Completion 2019-12 (Actual); Study Completion 2026-12-31 (Estimated)

PRIMARY OUTCOMES:
Cancer specific survival | 10 years
  Follow-up visits every 3 months

SECONDARY OUTCOMES:
Developement of castration-resistance measured by PSA value | 10 years
  Follow-up visits every 3 months
Overall survival | 10 years
  Follow-up visits every 3 months
Progression-free survival | 10 years
  Follow-up visits every 3 months

OTHER OUTCOMES:
Quality of Life measured by the EPIC-26 | 10 years
  Using a questionnaire, Follow-up visits every 3 months

CONTACTS AND LOCATIONS:
Overall Officials: Markus Graefen, Professor, Principal Investigator — Martini-Klinik am UKE GmbH
Locations (1):
- Markus Graefen, Hamburg, Nein, Germany

REFERENCES:
- [Background] Heidenreich A, Bastian PJ, Bellmunt J, Bolla M, Joniau S, van der Kwast T, Mason M, Matveev V, Wiegel T, Zattoni F, Mottet N; European Association of Urology. EAU guidelines on prostate cancer. part 1: screening, diagnosis, and local treatment with curative intent-update 2013. Eur Urol. 2014 Jan;65(1):124-37. doi: 10.1016/j.eururo.2013.09.046. Epub 2013 Oct 6. PMID 24207135
- [Background] Schellhammer PF, Venner P, Haas GP, Small EJ, Nieh PT, Seabaugh DR, Patterson AL, Klein E, Wajsman Z, Furr B, Chen Y, Kolvenbag GJ. Prostate specific antigen decreases after withdrawal of antiandrogen therapy with bicalutamide or flutamide in patients receiving combined androgen blockade. J Urol. 1997 May;157(5):1731-5. PMID 9112515
- [Background] Isbarn H, Huland H, Graefen M. Results of radical prostatectomy in newly diagnosed prostate cancer: long-term survival rates in locally advanced and high-risk cancers. Dtsch Arztebl Int. 2013 Jul;110(29-30):497-503. doi: 10.3238/arztebl.2013.0497. Epub 2013 Jul 22. PMID 24000298
- [Background] Engel J, Bastian PJ, Baur H, Beer V, Chaussy C, Gschwend JE, Oberneder R, Rothenberger KH, Stief CG, Holzel D. Survival benefit of radical prostatectomy in lymph node-positive patients with prostate cancer. Eur Urol. 2010 May;57(5):754-61. doi: 10.1016/j.eururo.2009.12.034. Epub 2010 Jan 20. PMID 20106588
- [Background] Steuber T, Budaus L, Walz J, Zorn KC, Schlomm T, Chun F, Ahyai S, Fisch M, Sauter G, Huland H, Graefen M, Haese A. Radical prostatectomy improves progression-free and cancer-specific survival in men with lymph node positive prostate cancer in the prostate-specific antigen era: a confirmatory study. BJU Int. 2011 Jun;107(11):1755-61. doi: 10.1111/j.1464-410X.2010.09730.x. Epub 2010 Oct 13. PMID 20942833
- [Background] Widmark A, Klepp O, Solberg A, Damber JE, Angelsen A, Fransson P, Lund JA, Tasdemir I, Hoyer M, Wiklund F, Fossa SD; Scandinavian Prostate Cancer Group Study 7; Swedish Association for Urological Oncology 3. Endocrine treatment, with or without radiotherapy, in locally advanced prostate cancer (SPCG-7/SFUO-3): an open randomised phase III trial. Lancet. 2009 Jan 24;373(9660):301-8. doi: 10.1016/S0140-6736(08)61815-2. Epub 2008 Dec 16. PMID 19091394
- [Background] Zelefsky MJ, Eastham JA, Cronin AM, Fuks Z, Zhang Z, Yamada Y, Vickers A, Scardino PT. Metastasis after radical prostatectomy or external beam radiotherapy for patients with clinically localized prostate cancer: a comparison of clinical cohorts adjusted for case mix. J Clin Oncol. 2010 Mar 20;28(9):1508-13. doi: 10.1200/JCO.2009.22.2265. Epub 2010 Feb 16. PMID 20159826
- [Background] Warde P, Mason M, Ding K, Kirkbride P, Brundage M, Cowan R, Gospodarowicz M, Sanders K, Kostashuk E, Swanson G, Barber J, Hiltz A, Parmar MK, Sathya J, Anderson J, Hayter C, Hetherington J, Sydes MR, Parulekar W; NCIC CTG PR.3/MRC UK PR07 investigators. Combined androgen deprivation therapy and radiation therapy for locally advanced prostate cancer: a randomised, phase 3 trial. Lancet. 2011 Dec 17;378(9809):2104-11. doi: 10.1016/S0140-6736(11)61095-7. Epub 2011 Nov 2. PMID 22056152
- [Background] Cooperberg MR, Vickers AJ, Broering JM, Carroll PR. Comparative risk-adjusted mortality outcomes after primary surgery, radiotherapy, or androgen-deprivation therapy for localized prostate cancer. Cancer. 2010 Nov 15;116(22):5226-34. doi: 10.1002/cncr.25456. PMID 20690197
- [Background] Wirth M, Tammela T, Cicalese V, Gomez Veiga F, Delaere K, Miller K, Tubaro A, Schulze M, Debruyne F, Huland H, Patel A, Lecouvet F, Caris C, Witjes W. Prevention of bone metastases in patients with high-risk nonmetastatic prostate cancer treated with zoledronic acid: efficacy and safety results of the Zometa European Study (ZEUS). Eur Urol. 2015 Mar;67(3):482-91. doi: 10.1016/j.eururo.2014.02.014. Epub 2014 Feb 20. PMID 24630685
- [Background] James ND, Sydes MR, Clarke NW, Mason MD, Dearnaley DP, Spears MR, Ritchie AW, Parker CC, Russell JM, Attard G, de Bono J, Cross W, Jones RJ, Thalmann G, Amos C, Matheson D, Millman R, Alzouebi M, Beesley S, Birtle AJ, Brock S, Cathomas R, Chakraborti P, Chowdhury S, Cook A, Elliott T, Gale J, Gibbs S, Graham JD, Hetherington J, Hughes R, Laing R, McKinna F, McLaren DB, O'Sullivan JM, Parikh O, Peedell C, Protheroe A, Robinson AJ, Srihari N, Srinivasan R, Staffurth J, Sundar S, Tolan S, Tsang D, Wagstaff J, Parmar MK; STAMPEDE investigators. Addition of docetaxel, zoledronic acid, or both to first-line long-term hormone therapy in prostate cancer (STAMPEDE): survival results from an adaptive, multiarm, multistage, platform randomised controlled trial. Lancet. 2016 Mar 19;387(10024):1163-77. doi: 10.1016/S0140-6736(15)01037-5. Epub 2015 Dec 21. PMID 26719232
- [Background] Sweeney CJ, Chen YH, Carducci M, Liu G, Jarrard DF, Eisenberger M, Wong YN, Hahn N, Kohli M, Cooney MM, Dreicer R, Vogelzang NJ, Picus J, Shevrin D, Hussain M, Garcia JA, DiPaola RS. Chemohormonal Therapy in Metastatic Hormone-Sensitive Prostate Cancer. N Engl J Med. 2015 Aug 20;373(8):737-46. doi: 10.1056/NEJMoa1503747. Epub 2015 Aug 5. PMID 26244877
- [Derived] Graefen M, Falkenbach F, Maurer T, Budaus L, Tilki D, Karakiewicz PI, Aly M, Wiklund P, Brasso K, Roder A, Poulsen MH, Schostak M, Gortzen C, Renter A, von Amsberg G, Haese A, Heinzer H, Salomon G, Steuber T, Beyer B. Best Systemic Therapy With or Without Radical Prostatectomy in the Management of Men With Oligometastatic Prostate Cancer: The RAMPP Randomised Controlled Trial. Eur Urol. 2025 Oct 3:S0302-2838(25)04687-1. doi: 10.1016/j.eururo.2025.09.4144. Online ahead of print. PMID 41046179